CLINICAL TRIAL: NCT06976021
Title: Immune PET and Proteomics for the Assessment of Response to Spatially Fractionated or Palliative Radiotherapy With or Without Immunotherapy Ocena Efektu immunomodulującego Radioterapii Paliatywnej, w Tym Radioterapii z Przestrzennym zróżnicowaniem Dawki, Podanej Samodzielnie Lub z immunoterapią, u Chorych którzy Wyczerpali możliwość Leczenia Systemowego i Radioterapii Radykalnej, Przy Wykorzystaniu Immuno-PET i badań Proteomicznych
Brief Title: Immune PET and Proteomics for the Assessment of Response to Spatially Fractionated or Palliative Radiotherapy With or Without Immunotherapy
Acronym: INTROSPECTION
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23/ABM/01/00078
Record Dates: First submitted 2025-04-27; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Triple Negative Breast Cancer; Uterine Cervical Cancer; Uterine Corpus Cancer; Malignant Melanoma; Clear Cell Renal Cell Carcinoma
Keywords: spatially fractionated radiotherapy; immunotherapy; immuno-PET; proteomics; signaling pathways
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Uterine Cervical Neoplasms; Melanoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SFRT with immunotherapy (Experimental)
  Interventions: Diagnostic Test: Baseline 89-Zr Pembrolizumab Immuno PET-CT; Diagnostic Test: Proteomic assay
- SHORT with immunotherapy (Active Comparator)
  Interventions: Diagnostic Test: Baseline 89-Zr Pembrolizumab Immuno PET-CT; Diagnostic Test: Proteomic assay
- SFRT (Experimental)
  Interventions: Diagnostic Test: Baseline 89-Zr Pembrolizumab Immuno PET-CT; Diagnostic Test: Proteomic assay; Diagnostic Test: Follow-up 89-Zr Pembrolizumab Immuno PET-CT
- SHORT (Active Comparator)
  Interventions: Diagnostic Test: Baseline 89-Zr Pembrolizumab Immuno PET-CT; Diagnostic Test: Proteomic assay; Diagnostic Test: Follow-up 89-Zr Pembrolizumab Immuno PET-CT

INTERVENTIONS:
Diagnostic Test: Baseline 89-Zr Pembrolizumab Immuno PET-CT — Diagnostic imaging with novel radiotracer - drug (Pembrolizumab) labeled with zirconium-89
Diagnostic Test: Proteomic assay — Assessment of the proteomic profile before and periodically after treatment
Diagnostic Test: Follow-up 89-Zr Pembrolizumab Immuno PET-CT — Diagnostic imaging with novel radiotracer - drug (Pembrolizumab) labeled with zirconium-89 after radiotherapy performed in patients who are not treated with immunotherapy
  Arms: SFRT; SHORT

SUMMARY:
The aim of the study is to evaluate the response to four schemes of treatment with novel diagnostic tools - Immuno-PET and proteomics as well as standard imaging (magnetic resonsonce imaging and computed tomography). Two fractionation schedules of radiotherapy will be used. The first will be a common standard of palliative irradiation - 20 Gy delivered in five fractions of 4 Gy (SHORT). The other is called Spatially Fractionated Radiotherapy (SFRT). SFRT is delivered in one fraction of 20 Gy but the dose is diversified inside the tumor to produce areas of high and low doses distributed alternately. This kind of irradiation may be able to stimulate immune response and improve the efficiency of immunotherapy. A drug belonging to the class of immunotherapeutic agents - Pembrolizumab will be added to the treatment scheme in two arms of the study to check that assumption. The response of the target tumor will be evaluated with PET study using Pembrolizumab labeled with zirconium-89 which will show the spatial distribution of immune receptors within the target tumor and other involved sites if there are any. The examination will be repeated after the treatment to evaluate changes in distribution of the immune receptors necessary for the drug to work. Additionally, the researchers will repeatedly test the presence and concentration of a wide panel of proteins in blood to evaluate response to the treatment more precisely.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of clear cell renal cell carcinoma, melanoma, cervical cancer, endometrial cancer or triple negative breast cancer.
2. Patients nnot eligible for radical treatment with radiotherapy (including stereotactic radiotherapy of the tumor in the potential planned area of irradiation in the study), chemotherapy and palliative immunotherapy in accordance with applicable national standards but who qualify for palliative radiation treatment
3. General condition according to Karnofsky scale: 60-100
4. Patients with tumor (index lesion) larger than 5 cm in size that can be irradiated with either SHORT or SFRT technique (presence of other tumors that may be independently treated locally is not an exclusion criterion)
5. The tumor may be assessed using iRECIST
6. Age over 18 years
7. Granted written, informed consent to participate in the research experiment
8. No contraindications to treatment with Pembrolizumab (according to the information provided in the product characteristics).
9. Expected survival time over 6 months.

Exclusion criteria

1. Lack of consent to participate in the experiment
2. Contraindications to Pembrolizumab according to the product characteristics
3. Pregnancy and lactation
4. Inability of the patient to cooperate, including claustrophobia that prevents imaging tests from being performed as planned.
5. Women of childbearing potential who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy throughout treatment and for 5 months after its completion.
6. Condition after organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in expression of PD-1 receptors expressed as a ratio of SUV values | one year
  The expression of PD-1 receptors will be measured with Immuno-PET basing on Zr-89 labeled Pembrolizumab and expressed as the ratio of initial and post-treatment SUV
Change in number of areas with PD-1 receptors expressed as number of lesions | one year
  The localization of regions expressing PD-1 receptors will be identified with Immuno-PET basing on Zr-89 labeled Pembrolizumab and expressed as the number of lesions
Change of proteome expression profile after treatment expressed in NPX (Normalized Protein eXpression) values | one year
  The difference between proteome expression profile before treatment and after the last infusion of Pembrolizumab or after a year in arms without immunotherapy. The Proximity Extension Assay (PEA) technology will be used. Following sequencing, the raw data will be converted to counts, assigning an integer value to each assay-sample combination based on the detected copy numbers. These raw data counts will be converted into NPX values, enabling the identification of protein level changes within different sample sets, and establishing protein signatures.

CONTACTS AND LOCATIONS:
Overall Officials: Sławomir Blamek, MD, PhD, MBA, Principal Investigator — Maria Skłodowska-Curie National Research Institute of Oncology, Gliwice Branch

IPD SHARING:
Plan to Share IPD: Yes
The individual patient data can be shared upon request. The basic demographic data, type of intervention and outcome measures will be available.
Supporting Information: Study Protocol, ICF, CSR